CLINICAL TRIAL: NCT04540406
Title: Modulation of Gut Microbiota With NBT-NM108 as an Early Treatment for Suspected or Confirmed Symptomatic COVID-19 Patients
Brief Title: NBT-NM108 as an Early Treatment for Suspected or Confirmed Symptomatic COVID-19 Patients
Acronym: COVGUT20
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Notitia Biotechnologies Company (Industry)
Collaborators: University of South Florida (Other); Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBTNM10810012020
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Suspected or Confirmed COVID-19
Keywords: COVID-19; NBT-NM108; Notitia Biotechnologies Company; Notitia Biotechnologies; Microbiome; Microbiota; Gut microbiome; Gut microbiota; Corona Virus; Novel Corona Virus; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBT-NM108 + Usual Care (Experimental)
  Interventions: Drug: NBT-NM108
- Usual Care Only (Active Comparator)
  Interventions: Other: Usual Care Only

INTERVENTIONS:
Drug: NBT-NM108 — Taken in the form of drinks four times a day (before each main meal and 2 hours after dinner) for 28 days. Each drink is prepared by mixing one sachet (30 g) with 500 ml of water.
  Arms: NBT-NM108 + Usual Care
Other: Usual Care Only — Control group will also follow the same schedule except they will drink the same volume of water without NBT-NM108.
  Arms: Usual Care Only

SUMMARY:
This open-label, randomized, and controlled clinical trial aims to determine the feasibility and effectiveness of using NBT-NM108, a novel botanical-based fixed-combination drug, to modulate the gut microbiota and treat early-stage suspected or confirmed symptomatic COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 79 (inclusive)
* Have mild to moderate COVID-19-like symptoms based on the symptom list from CDC (updated May 13, 2020) and the severity categorization from FDA [18]:

  a) Mild COVID-19
* Fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, and diarrhea
* No clinical signs indicative of moderate, severe, or critical illness severity

  b) Moderate COVID-19
* Symptoms of moderate illness with COVID-19 could include any symptom of mild illness or shortness of breath with exertion
* Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≥ 20 breaths/min, oxygen saturation level > 93% on room air at sea level, heart rate ≥ 90 beats/min
* No clinical signs indicative of severe or critical illness severity
* Directed to home isolation by study physician
* Confirm study enrollment within 7 days of symptom onset
* Practice acceptable contraception, i.e., continue with current methods if participants are already practicing contraception, otherwise participants must agree to practicing contraception with a barrier method (male or female condom) or abstinence, from Day 1 to Day 35 or 7 days after the last dose of NBT-NM108 if they do not complete the 28-day intervention.
* Have access to a smartphone, tablet, computer, or other qualifying internet-enabled device and daily internet access
* Understand and be able to follow written and oral instructions in English
* Provide informed consent

Exclusion Criteria

* Have tested positive for COVID-19 and recovered
* Receiving vancomycin monotherapy or oral broad-spectrum antibiotics
* Inability to receive oral fluids
* Self-reported allergy or intolerance to any ingredients in NBT-NM108
* Surgery involving the intestinal lumen within the last 30 days
* Documented diagnosis of celiac disease, inflammatory bowel disease or irritable bowel syndrome
* Pregnancy or breastfeeding
* Bariatric surgery
* Immunocompromised, e.g., cancer treatment, bone marrow/organ transplant, immune deficiency, poorly controlled HIV/AIDS, prolonged use of steroids or other immunosuppressant medications

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asa Oxner, MD, Principal Investigator — University of South Florida; Liping Zhao, PhD, Principal Investigator — Rutgers University
Locations (1):
- University of South Florida Morsani College of Medicine, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Started | 23 | 19
Completed | 16 | 15
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (11.4) | 45.7 (10.1) | 44.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Amplicon Sequence Variants (ASVs) That Are Significantly Correlated With Variation in the Microbiome Data Between NBT-NM108 Group and Usual Care Only Group From Day 0 to 28
Description: Amplicon Sequence Variants (ASVs) significantly correlated with the first principal coordinate (PC1) from the covariate-adjusted Principal Coordinates Analysis (aPCoA) were identified, each having an average relative abundance greater than 0.001%. These ASVs represent specific microbial features whose relative abundance was most strongly associated with the primary axis of variation in the microbiome data, after adjusting for covariates. It was hypothesized that PC1 might reflect the direction of microbiome changes induced by the intervention, given its association with shifts observed in participants' microbiome compositions before and after the intervention. The unit of measure used here is the relative abundance percentage of each ASV in the stool sample.
Time Frame: Day 0-28
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- NBT-NM108 + Usual Care (Day 0); NBT-NM108 + Usual Care (Day 28): NBT-NM108: Taken in the form of drinks four times a day (before each main meal and 2 hours after dinner) for 28 days. Each drink is prepared by mixing one sachet (30 g) with 500 ml of water.
- Usual Care Only (Day 0); Usual Care Only (Day 28): Usual Care Only: Control group will also follow the same schedule except they will drink the same volume of water without NBT-NM108.
Arm/Group | NBT-NM108 + Usual Care (Day 0) | Usual Care Only (Day 0) | NBT-NM108 + Usual Care (Day 28) | Usual Care Only (Day 28)
Number analyzed (Participants) | 16 | 15 | 16 | 15
percentage
  Agathobacter ASV00LE (positively correlated with PC1) | 7.74 (8.227) | 6.251 (7.363) | 7.986 (7.997) | 5.54 (5.399)
  Roseburia ASV01JE (negatively correlated with PC1) | 1.211 (2.551) | 0.857 (1.031) | 0.703 (0.77) | 1.054 (1.23)
  Lachnoclostridium ASV0034 (negatively correlated with PC1) | 0.13 (0.153) | 0.164 (0.149) | 0.185 (0.273) | 0.142 (0.198)
  Fusicatenibacter ASV07L5 (negatively correlated with PC1) | 0.092 (0.201) | 0.23 (0.457) | 0.067 (0.191) | 0.122 (0.252)
  Bacteroides_uniformis ASV04EI (negatively correlated with PC1) | 0.096 (0.364) | 0.044 (0.181) | 0.311 (1.131) | 0.043 (0.168)
  Phascolarctobacterium ASV0EJD (negatively correlated with PC1) | 0.154 (0.597) | 0.068 (0.279) | 0.225 (0.98) | 0.072 (0.279)
  Veillonella ASV0065 (negatively correlated with PC1) | 0.022 (0.048) | 0.1 (0.246) | 0.029 (0.089) | 0.088 (0.228)
  Lachnospiraceae ASV030X (negatively correlated with PC1) | 0.019 (0.035) | 0.02 (0.046) | 0.024 (0.065) | 0.02 (0.041)
  Shuttleworthia ASV03B1 (negatively correlated with PC1) | 0.014 (0.059) | 0.012 (0.025) | 0.004 (0.013) | 0.007 (0.019)
  Parabacteroides ASV000W (negatively correlated with PC1) | 0.003 (0.013) | 0 (0) | 0.01 (0.042) | 0 (0)
  Lachnoclostridium ASV0055 (negatively correlated with PC1) | 0.005 (0.023) | 0.009 (0.025) | 0.006 (0.024) | 0 (0)
  Lachnospiraceae ASV05T7 (negatively correlated with PC1) | 0.001 (0.004) | 0.005 (0.011) | 0.001 (0.003) | 0.002 (0.006)
  Ruminococcus_gauvreauii_group ASV0GHA (negatively correlated with PC1) | 0.002 (0.012) | 0 (0) | 0.003 (0.013) | 0 (0)
  Lachnospiraceae_NK4A136_group ASV0GHH (negatively correlated with PC1) | 0.004 (0.022) | 0 (0) | 0.001 (0.004) | 0 (0)
  Acetanaerobacterium ASV00E7 (negatively correlated with PC1) | 0.002 (0.004) | 0.001 (0.003) | 0.001 (0.003) | 0.001 (0.003)
  Lachnospiraceae ASV0074 (negatively correlated with PC1) | 0.003 (0.009) | 0.001 (0.005) | 0.002 (0.006) | 0 (0)
  Eggerthellaceae ASV0G1P (negatively correlated with PC1) | 0.001 (0.002) | 0.003 (0.007) | 0 (0.001) | 0.002 (0.003)
  Lachnospiraceae_UGG-010 ASV06Y8 (negatively correlated with PC1) | 0.002 (0.005) | 0 (0) | 0.004 (0.014) | 0 (0)
  Lachnospiraceae_GCA_900066575 ASV03BI (negatively correlated with PC1) | 0 (0.001) | 0.001 (0.003) | 0 (0.002) | 0.002 (0.006)
  Frisingicoccus ASV0EAB (negatively correlated with PC1) | 0.001 (0.005) | 0 (0) | 0 (0.002) | 0 (0)
Statistical Analysis 1: Comparison: Usual Care Only (Day 0) vs Usual Care Only (Day 28); PCoA (Principal Coordinates Analysis) + PERMANOVA (Permutational Multivariate Analysis of Variance) are exploratory multivariate techniques commonly used in microbiome research to assess and visualize differences in community composition. The null hypothesis for PERMANOVA is that there are no differences in the centroids (multivariate means) of the groups being compared. The microbial communities in different groups or conditions are not significantly different from each other; Test type: Other — We employed covariate-adjusted Principal Coordinates Analysis and a subject-stratified PERMANOVA test to assess the overall gut microbiota structural change. These tests are generally neither superiority, non-inferiority, nor equivalence tests. Instead, they are used to detect and evaluate overall differences in the microbial community structure between groups or conditions; To assess the overall structural changes in gut microbiota, we employed covariate-adjusted Principal Coordinates Analysis (PCoA) and a subject-stratified PERMANOVA test. PCoA, an exploratory multivariate technique, helps visualize and interpret patterns in complex microbiome data by reducing dimensionality, with the first principal coordinate (PC1) capturing the largest variation among samples. PERMANOVA, which does not rely on standard parametric assumptions, was used to determine if there are statistically significant differences in the overall composition of microbial communities between groups based on a chosen distance metric. Our analysis aimed to explore whether microbial community compositions differed significantly between Day 0 and Day 28 within the Treatment group, accounting for inter-individual variability. Similarly, we investigated if such differences existed over the same time points in the Control group. The unit of measure was distance metrics

2. Secondary Outcome: Number of Participants That Were Hospitalized or Died From COVID19
Description: Hospitalization or death
Time Frame: At days 0, 14, 28, and 56
Measure: Count of Participants; unit: Participants
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Participants
  Day 0 | 0 | 0
  Day 14 | 0 | 0
  Day 28 | 0 | 0
  Day 56 | 0 | 0

3. Secondary Outcome: Proportion of Participants Who Are "Alive and Not Admitted to the Hospital"
Description: (not specified)
Time Frame: At days 0, 14, 28, and 56
Measure: Count of Participants; unit: Participants
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Participants
  Day 0 | 16 | 15
  Day 14 | 16 | 15
  Day 28 | 16 | 15
  Day 56 | 16 | 15

4. Secondary Outcome: Number of Participants Who Visited the Emergency Room From COVID-19
Time Frame: At days 0, 14, 28, and 56
Measure: Count of Participants; unit: Participants
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Participants
  Day 0 | 0 | 0
  Day 14 | 0 | 0
  Day 28 | 0 | 0
  Day 56 | 0 | 0

5. Secondary Outcome: Proportion of Participants Who Have Complete Resolution of Objective Symptoms
Description: All vitals signs are within normal range for at least 24h, including body temperature 36.4-37.5C (97.7-99.5F), pulse rate <90/min, respiratory rate 12-16/min, and oxygen saturation level at 95-100%.
Time Frame: At days 28 and 56
Measure: Count of Participants; unit: Participants
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Participants
  Day 28 | 11 | 11
  Day 56 | 16 | 15

6. Secondary Outcome: Proportion of Participants Who Have Complete Resolution of Subjective Symptoms
Description: Absence of all COVID-19-like symptoms listed by CDC (updated May 13, 2020) for at least 48h, including the presence of chills or "feeling feverish" , cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting and diarrhea
Time Frame: At days 28 and 56
Measure: Count of Participants; unit: Participants
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Participants
  Day 28 | 5 | 7
  Day 56 | 16 | 15

7. Secondary Outcome: Proportion of Participants Who Have Complete Resolution of Subjective Symptoms Except Fatigue and Cough
Description: Proportion of participants who have complete resolution of subjective symptoms except fatigue and cough, i.e. absence of all COVID-19-like symptoms listed by CDC (updated May 13, 2020) for at least 48 h, including the presence of chills or "feeling feverish", cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting and diarrhea
Time Frame: At days 28 and 56
Measure: Count of Participants; unit: Participants
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Participants
  Day 28 | 5 | 7
  Day 56 | 16 | 15

8. Secondary Outcome: Illness Severity Based on the Categorization From FDA and World Health Organization COVID-19 Guidance Document
Description: Proportion of participants who meet each COVID-19 category in both mild, moderate, and severe categories
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Participants
  mild | 8 | 7
  moderate | 8 | 8
  severe | 0 | 0

9. Secondary Outcome: Oral Body Temperature (F)
Time Frame: At days 0, 14, 28, and 56
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit (F)
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
Degrees Fahrenheit (F)
  Day 0 | 97.1 (1.2) | 97.4 (1.3)
  Day 14 | 97.9 (0.5) | 97.3 (0.6)
  Day 28 | 97.1 (0.8) | 97.4 (0.7)
  Day 56 | 97.6 (1.0) | 97.1 (0.9)

10. Secondary Outcome: Oxygen Saturation SpO2 Level
Time Frame: At days 0, 14, 28, and 56
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
percentage of oxygen saturation
  Day 0 | 96.5 (1.7) | 97.3 (1.3)
  Day 14 | 98.1 (1.1) | 97.6 (1.0)
  Day 28 | 97.0 (1.2) | 98.4 (1.1)
  Day 56 | 93.0 (1.1) | 94.0 (1.2)

11. Secondary Outcome: Pulse Rate Per Minute
Time Frame: At days 0, 14, 28, and 56
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
beats per minute
  Day 0 | 78.0 (9) | 79.9 (10.1)
  Day 14 | 79.7 (5.9) | 78.8 (6.2)
  Day 28 | 71.0 (6.5) | 72.1 (9.4)
  Day 56 | 70.5 (6.7) | 71 (6.3)

12. Secondary Outcome: Respiratory Rate Per Minute
Time Frame: At days 0, 14, 28, and 56
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
breaths per minute
  Day 0 | 18.1 (12.1) | 18.3 (13.2)
  Day 14 | 17.0 (5.0) | 17.5 (4.5)
  Day 28 | 15.4 (4.9) | 14.1 (5.1)
  Day 56 | 13.6 (5.0) | 14 (5.2)

13. Secondary Outcome: Fasting Blood Glucose
Time Frame: At days 0 and 28
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
Number analyzed (Participants) | 16 | 15
mg/dL
  Day 0 | 91 (6) | 92 (6.8)
  Day 28 | 90 (5.2) | 89 (7)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | NBT-NM108 + Usual Care | Usual Care Only
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 3/16 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBT-NM108 + Usual Care (N=16) | Usual Care Only (N=15)
Mild adverse events (General disorders) | 3 (3) | 0 (0) — mild adverse events include bloating, abdominal discomfort, and Pruritus

LIMITATIONS AND CAVEATS:
The primary limitation of our randomized controlled trial is the restriction of our study population to patients with mild to moderate COVID-19. Consequently, the findings may not be generalizable to individuals with severe or critical COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT04540406/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT04540406/SAP_001.pdf